CLINICAL TRIAL: NCT06205303
Title: An Interventional Study to Improve Medication Adherence Using Patient Decision Aid Among Adults With Under-Replaced HypoThyroidism (IMPART): A Randomized Control Study
Brief Title: Interventional Study to Improve Medication Adherence Using Patient Decision Aid
Acronym: IMPART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SingHealth Polyclinics (Other)
Responsible Party: Principal Investigator, Kalaipriya Gunasekaran, Principal Investigator, SingHealth Polyclinics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/2466
Record Dates: First submitted 2023-12-27; First posted 2024-01-16 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hypothyroidism
Keywords: thyroxine; under-replacement; medication adherence; PDA; intervention
MeSH Terms: conditions — Hypothyroidism; Medication Adherence | interventions — Videotape Recording

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm using PDA (Experimental): The intervention arm participants will watch the PDA which is estimated to take 10 minutes, after their consultation with the physician. The participants will be directed to a private room to watch the PDA.
  Interventions: Other: Patient Decision Aid (Video)
- Control arm (No Intervention): The control arm participants will receive a thyroxine replacement pamphlet at their routine clinic appointment but will not attend the health education session using the PDA.

INTERVENTIONS:
Other: Patient Decision Aid (Video) — Patient decision aid on thyroxine replacement is a video designed to assist the hypothyroid adults with under-replacement. It provides clear and balanced information about hypothyroidism, the role of thyroxine, treatment benefits, potential risks, and factors interfering thyroxine absorption and bioavailability. The PDA aims to empower patients to engage in shared decision-making with their healthcare provider, ensuring they understand the options and can make choices aligned with their preferences and values.
  Arms: intervention arm using PDA

SUMMARY:
Background:

Although hypothyroidism is easily treated with levothyroxine (LT4) replacement, results from several studies indicate that people receiving LT4 replacement often have under- or over-replaced thyroid function. Poor medication adherence and factors interfering with thyroxine absorption and bioavailability may result in such under-replacement. Using the COM-B (Capability, Motivation, and Opportunity - Behavior) model, a health education intervention using patient decision aid (PDA), was developed for primary care physicians to educate individuals about thyroxine replacement. Besides imparting health literacy, PDAs provide greater comfort of the patients to participate in decision making. Intervention with the PDA aims to improve the medication adherence by increasing patients' knowledge about thyroxine replacement.

Specific aims: The primary aim is to determine effectiveness of PDA in improving the knowledge, medication adherence and quality of life of the under-replaced hypothyroid adults in a primary care setting. Secondary aims are to explore their understanding and acceptance on the PDA and to assess their perceived usability of this PDA.

Methodology: A randomised controlled trial will be conducted at SingHealth Polyclinics (SHP) using mixed-method study design to determine effectiveness of PDA. Patient participants will be randomly allocated in a 1:1 ratio to either the intervention or control group. A total of 236 (118 in each group) patient participants will be enrolled by simple randomization. Eligible patient must be of age ≥21 years years and have LT4 under-replacement with Thyroid stimulating hormone (TSH) >3.7 mIU/L within the last 6 months.

Relevance/significance of the study: Findings from the study may add evidence to the scientific knowledge of using PDA to improve medication adherence and recommend development of similar interventions for other chronic medical conditions.

DETAILED DESCRIPTION:
Patient decision aids (PDA) help people involved in decision making by providing information about the options and outcomes, and by clarifying their concerns. PDAs will help the patients to participate in decision making through SHARE approach (seeking patients' participation, helping them to explore and compare treatment options, assessing their values and preferences, reaching a decision with them and evaluating the patients' decision). Decision aids have the potential to improve adherence by enabling patient-doctor communication on treatment-related factors.

PDAs have been shown to improve medication adherence across different chronic diseases like osteoporosis and prevention of coronary heart diseases with aspirin. These aids provide patients with valuable information and support, helping them make informed choices about their treatment plans and fostering better adherence to prescribed medications. Decision Aids are available for managing hyperthyroidism caused by Grave's disease, but not for hypothyroidism. Addressing this gap could greatly empower patients with hypothyroidism to make well-informed choices about their treatment and improve their overall experience with managing this condition.

Intervention and theoretical framework According to the Capability, Motivation, and Opportunity - Behavior (COM-B) model, Capability, Motivation, and Opportunity are all referred to as "components" that influence behavior. Capability refers to the 'individual's psychological and physical capacity to engage in the activity concerned' while Opportunity refers to all those 'factors that lie outside the individual that make the behaviour possible or provoke it.' Motivation includes 'all those cognitive processes that motivate direct behavior including the habitual processes, emotional responding and analytical decision-making.' Earlier models to improve medication adherence generally highlighted the importance of doctor-patient communication and its impact on patient satisfaction, knowledge and ignorance as key determinants of medication adherence. However, studies on health behavior have constantly shown that merely providing information alone is not an effective strategy to influence behavior like adherence to medication. The COM-B model explicitly considers external resources like physical and social environment, which are typically not considered in other models like transtheoretical model of behavior change or health belief model. Jackson et al considered that COM-B model provided a more comprehensive description of adherence than other existing models, making it easier to identify appropriate interventions.

Study objectives The aim is to evaluate the acceptance, usability, understanding and effectiveness of a PDA developed for hypothyroid adults in improving their knowledge, beliefs, adherence and quality of life in patients with under-replaced hypothyroid status in primary care.

Primary objective is

• To determine effectiveness of PDA in improving the knowledge, beliefs, medication adherence and quality of life

Secondary objectives are as follows:

i) To assess their perceived usability of this PDA ii) To assess patients' understanding and acceptance on the PDA

Recruitment and consent taking Participant recruitment Eligible patient participants will be referred by the attending physicians to the study team. The study team will verify eligibility of shortlisted patients using an eligibility assessment form and written informed consent will be obtained in-person at the study site, in a quiet and separate room or space free from intrusion. The participant will sign three hardcopies of the consent form. One copy each will be kept by the participant, study team and the participants' electronic medical records. Adequate time will be given to read the documents and to ask any questions. Assurance will be given that the decision whether to participate is entirely voluntary and will not result in any compromise of their routine clinical care.

Participant withdrawal Participants may choose to withdraw from the study at any time without providing an explanation and this will not result in any punitive consequences.

Randomization Participants will be randomized to either the intervention arm (health education using the PDA) or the control arm (thyroxine replacement pamphlet during routine clinic appointment) in a ratio of 1:1, using computer-generated random numbers for simple randomization of subjects. Patient participants will not be blinded to the allocation status. The randomization sequence is written and kept in an opaque sealed envelope, which will be labelled with a serial number. The study team will open the sealed envelope once the patient has consented to participate and then will be assigned to the intervention arm accordingly.

Blinding The nature of the intervention makes impossible to blind patients and research team to participant allocation. However, treating doctors will be blinded to the allocated group as the intervention session using the PDA will be delivered after their routine clinic appointment and dose titration, if required. The data analysts will also be blinded to the allocated group before analysis.

Follow-up The primary goal of thyroxine replacement is to maintain thyroid hormone levels within a normal range. Since TSH responds sensitively to these levels (free T4/T3), clinical practice guidelines recommend using TSH levels as the primary marker for monitoring thyroxine replacement. Hence only TSH will be used to monitor the participants.

ELIGIBILITY:
Inclusion criteria

* Age ≥21 years
* Able to read and speak English
* Active patient with hypothyroidism at SingHealth Polyclinics (SHP) {had minimum of 2 follow-up visits at the respective study site in the last 12 months}
* TSH >3.70 milli-international units per liter (mIU/L)

Exclusion Criteria:

* Euthyroid state (TSH 0.65-3.70 mIU/L)
* LT4 over-replacement (TSH <0.65 mIU/L)
* Individuals who are severely ill or with hearing impairment and mental disturbances
* Pregnant women
* Sick euthyroid syndrome

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge about thyroxine replacement | through study completion, an average of 8 weeks to 9 months
  Change in the scores using knowledge on thyroxine replacement questionnaire; a newly developed knowledge questionnaire to access patients' understanding of thyroxine replacement comprising 16 questions scored from a scale of 0-5: 0 (Always), 1 (a few times a week), 2 (once a week or less), 3 (a few times a month), 4 (once a month or less) and 5 (Never). A higher score indicates better understanding.
Medication adherence | through study completion, an average of 8 weeks to 9 months
  Change in the scores using five-item Medication Adherence Report Scale (MARS-5); MARS-5 score was calculated by summing the numeric score (range 1-5) from each question for out of 25 (range 5-25). A higher score indicates better adherence.
Beliefs about medication | through study completion, an average of 8 weeks to 9 months
  Change in the scores using Beliefs About Medicines Questionnaire (BMQ). The BMQ is an 18-item questionnaire which consists of two components assessing patient's perceptions towards medications, BMQ-Specific and BMQ-General. The responses in both subscales are recorded on a five-point Likert scale. A higher score indicate stronger beliefs.
Health related Quality of life | through study completion, an average of 8 weeks to 9 months
  Change in the scores using the 5 Level EuroQol-5 Dimension (EQ-5D-5L) questionnaire; The EQ-5D-5L tool comprises five dimensions, each describing a different aspect of health: mobility, self-care, usual activities, pain/ discomfort and anxiety/ depression. Each dimension has five response levels (no problems, slight problems, moderate problems, severe problems, unable to/extreme problems). The proportion of patients reporting each level of problem on each dimension of the EuroQol-5 Dimension (EQ-5D) will be determined through study completion and compared. EuroQol Visual Analogue Scale (EQ VAS) provides a quantitative measure of the patient's perception of their overall health. The EQ VAS records the respondent's overall current health on a vertical scale (0-100), where the endpoints are labelled '0-The worst health you can imagine' and '100-The best health you can imagine'.

SECONDARY OUTCOMES:
Usability of PDA | after the intervention up to 9 months
  Measured using system usability scale (SUS). The SUS had 10 statements, and a 5-point Likert scale was used to indicate the participant's agreement with the statements. The mean score was calculated from the intervention group and a SUS score above 68 would be considered above average and anything below 68 is below average in terms of usability.
Patients' understanding and acceptance | immediately after the intervention
  in-depth interview with the participants in intervention arm till point of data saturation

CONTACTS AND LOCATIONS:
Overall Officials: Kalaipriya Gunasekaran, MD, Principal Investigator — SingHealth Polyclinics
Locations (1):
- SingHealth Polyclinics, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tan NC, Chew RQ, Koh YLE, Subramanian RC, Sankari U, Meyappan M, Cho LW. Primary hypothyroidism in the community: Lower daily dosages of levothyroxine replacement therapy for Asian patients. Medicine (Baltimore). 2017 Feb;96(7):e6145. doi: 10.1097/MD.0000000000006145. PMID 28207545
- [Background] Crilly M, Esmail A. Randomised controlled trial of a hypothyroid educational booklet to improve thyroxine adherence. Br J Gen Pract. 2005 May;55(514):362-8. PMID 15904555
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Jackson C, Eliasson L, Barber N, Weinman J. Applying COM-B to medication adherence: a suggested framework for research and interventions. Eur Health Psychol. 2014;16:7-17.